CLINICAL TRIAL: NCT02290860
Title: Screening Type 2 Diabetes Mellitus on the 2nd Day After Delivery in Women With Gestational Diabetes Mellitus - Stage 2, a Multicentre Trial.
Brief Title: Screening Type 2 Diabetes Mellitus on the 2nd Day After Delivery in Women With Gestational Diabetes Mellitus
Acronym: SoL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: University of Toronto (Other); University of Manitoba (Other)
Responsible Party: Principal Investigator, Jean-Luc Ardilouze, Endocrinologist, researcher, Université de Sherbrooke
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-161
Record Dates: First submitted 2014-11-10; First posted 2014-11-14 (Estimated); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Diabetes, Gestational
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Other): Type 2 diabetes diagnosis test.
  Interventions: Procedure: Type 2 diabetes diagnosis test

INTERVENTIONS:
Procedure: Type 2 diabetes diagnosis test — Participants will perform type 2 diabetes diagnosis test the day of hospital discharge after delivery and the same test around 8 weeks later.

SUMMARY:
Gestational diabetes mellitus (GDM) is defined as a hyperglycemia with onset or first recognition during pregnancy. GDM complicates 5 to 25% of pregnancies, depending on the diagnostic criteria used and the population being studied.

GDM is an important red flag: up to 70% women with GDM will develop type 2 diabetes mellitus (T2DM) during their lifetime. Accordingly, professional associations recommend T2DM postpartum screening (T2DM-pP-S), 6-to-24 weeks after delivery. A 75g oral glucose tolerance test (OGTT) should be performed for diagnosis (gold standard). Nevertheless, this T2DM-pP-S recommendation has failed worldwide for the same reasons: the presently impractical pattern of the testing. A solution is direly needed.

Our overall goal is to improve detection of pre-diabetes and diabetes and more specifically, to facilitate the recommended T2DM-pP-S in women diagnosed with GDM.

We hypothesize that, in GDM women, results of an OGTT performed after delivery, before hospital discharge (OGTT-1) predict results of the recommended OGTT at 6-to-12 weeks postpartum (OGTT-2). Our aims are:

1. To validate in Caucasian women the predictive threshold value of the 2hr-glucose of OGTT-1 established by our Stage-1 study.
2. To determine, in a multiethnic non-Caucasian cohort, the threshold value for the 2hr-glucose of OGTT-1 that is predictive of abnormal glucose tolerance at OGTT-2.
3. To define the OGTT time preference of women (before hospital discharge vs. 6-to-12 weeks postpartum).

If our results are in line with our Stage-1 data, most redundant 6-to-24 weeks postpartum OGTT will be avoided. Medical practice will change.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 18 and 45 years;
* Having a positive diagnosis of gestational diabetes mellitus (GDM) (IADPSG or CDA criteria or patient followed for GDM);
* Treated with diet, insulin or oral hypoglycemic agents;
* Have given birth to a child at term (gestational age ≥ 37 weeks);
* Have signed the consent form.

Exclusion Criteria:

* History of glucose intolerance or diabetes before the pregnancy;
* Have presented another obstetrical pathology during the pregnancy;

  * Severe gestational high blood pressure with proteinuria;
  * Delayed intrauterine development syndrome;
  * Pregnancy with more than a foetus;
  * Drug addiction;
  * Had complications during the delivery such as:
* Moderate to severe postpartum bleeding;
* Surgery in postpartum (curettage, hysterectomy, etc.).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 228 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
abnormal glucose tolerance | 8 weeks after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc Ardilouze, MD, PhD, Principal Investigator — Centre de recherche du Centre hospitalier universitaire de Sherbrooke
Locations (1):
- Centre de recherche clinique du CHUS, Sherbrooke, Quebec, Canada